CLINICAL TRIAL: NCT02433223
Title: Retrospective Evaluation of COPD Patient Care
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Queen Elizabeth Hospital (Other)
Responsible Party: Principal Investigator, Kristin Carson, Senior Research Scientist, The Queen Elizabeth Hospital
Other Study IDs: QElizabethH COPD
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: outreach nursing; respiratory nursing guidelines
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 2006 Patients: Comparison of Respiratory Chronic Disease Management provided against recommendations in 2005 Respiratory Nursing Guidelines through documentation
- 2011 Patients: Comparison of Respiratory Chronic Disease Management provided against recommendations in 2005 Respiratory Nursing Guidelines through documentation. With comparison of data against 2006 results.
- 2013 Patients: Comparison of Respiratory Chronic Disease Management provided against recommendations in 2005 Respiratory Nursing Guidelines through documentation. With comparison of data against 2006 & 2011 results.
- 2015 Patients: Group added to reflect recency of practice. Comparison of Respiratory Chronic Disease Management provided against recommendations in 2005 Respiratory Nursing Guidelines through documentation. With comparison of data against 2006 & 2011 results.

SUMMARY:
The purpose of this project is to evaluate hospital utilisation, patient and service outcomes of a Respiratory Nursing Service to examine current clinical care of COPD. This evaluation aims to identify the important gaps in current clinical care of respiratory chronic disease nursing management. The primary outcomes of this evaluation is to determine the efficacy of clinical care in 2006, 2011, 2013 and 2015 and compare data to current Nursing Best practice guidelines for COPD through the quantification of hospital utilisation for hospital admission, average length of stay, readmission within 28 days, emergency service attendance, outpatient review, use of Hospital and Home (H@H), frequency of exacerbations, disease severity and progression (FEV1: GOLD Classification), number of contacts with the respiratory nursing service and type of contacts with the respiratory nursing service.

DETAILED DESCRIPTION:
Study design: This study is a retrospective observational crosssectional study conducted through review of medical records, internal respiratory databases and electronic hospital patient record (OACIS & HOMER) over 3x12 blocks.

Participants: COPD patients from The Queen Elizabeth Hospital(TQEH) Respiratory Nursing Service who were new patients in 2006, 2011, 2013 and 2015 (Jan 1st to Dec 31st ). Data collection: Demographics, clinical data, hospital service utilisation, and clinical outcomes such as exacerbation frequency and disease progression. All data will be extracted into a standardised data extraction form, which a random subset will be checked by a second researcher.

Demographic data will include comparison of % without comorbidities, impact of comorbid conditions using Charleston Comorbidity index isolating diabetes, heart failure, anxiety and depression. Demographic and descriptive data will be given in means + SD and compared using a two-tailed Student t-test. Categorical variables will be compared using chisquared or Fisher exact tests, and when appropriate the MannWhitney Utest for nonparametric data. Statistical significance will be determined using an alpha of p <0.05. All analyses will be examined using SPSS software (version x).

ELIGIBILITY:
Inclusion Criteria

* any new client or new referral to the Respiratory Nursing Service in the years 2006, 2011, 2013 or 2015 only
* have a diagnosis of Chronic Obstructive Pulmonary Disease

Exclusion Criteria

* not a pre- existing client of the Respiratory Nursing Service
* not having a diagnosis of Chronic Obstructive Pulmonary Disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: New patients to the Respiratory Nursing Service in 2006, 2011, 2013 & 2015 with a diagnosis of Chronic Obstructive Pulmonary Disease
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of care provided by the Respiratory Nursing Service | 12 months
  Compare documentation against the components of 'Nursing Best Practice Guideline, Nursing Care of Dyspnea: The 6th Vital Sign in Individuals with Chronic Obstructive Pulmonary Disease (COPD)'

SECONDARY OUTCOMES:
Impact of respiratory nursing outreach on hospital, patient and service outcomes | 12 months
  Hospital utilisation is determined by hospital admissions, emergency department presentations, length of stay, readmission within 28 days, number of Respiratory Outpatient reviews and use of Hospital at Home. Patient outcomes are frequency of exacerbations, disease severity and progression (FEV1: GOLD Classification), Quality of Life, lung function and exercise tolerance. Respiratory Nurse outcomes are the number and type of contacts performed
Comorbidity in respiratory nursing | 12 months
  Identify the percentage of patients involved in the Respiratory Nursing Service with COPD who do and do not have a co-morbidity? Identify those with a comorbidity are they Aboriginal and Torres Strait Islander, of Cultural and Linguistic descent or of a low socioeconomic group? Identify the impact of co-morbid conditions using Charlson Comorbidity index isolating diabetes, heart failure, anxiety and depression?

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Smith, PhD, Study Director — The Queen Elizabeth Hospital

IPD SHARING:
Plan to Share IPD: Yes
Available upon request
Time Frame: Data analysis is expected to be completed by 30 June 2018
Access Criteria: For publication in nursing journal Sharing of information captured as requested